CLINICAL TRIAL: NCT04417894
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel- Group Study to Evaluate the Efficacy and Safety of Dupilumab in Adult and Adolescent Patients With Moderate-to-Severe Atopic Hand and Foot Dermatitis
Brief Title: A Study to Evaluate the Efficacy and Safety of Dupilumab in Adult and Adolescent Patients With Moderate-to-Severe Atopic Hand and Foot Dermatitis (Liberty-AD-HAFT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R668-AD-1924; 2019-003088-22 (EudraCT Number)
Record Dates: First submitted 2020-06-02; First posted 2020-06-05 (Actual); Results first posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Moderate to Severe Atopic Hand and Foot Dermatitis
MeSH Terms: interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- dupilumab (Experimental): Administered subcutaneously (SC) once every 2 weeks (Q2W), following a loading dose on Day 1
  Interventions: Drug: dupilumab
- Matching Placebo (Experimental): Administered SC Q2W, following a loading dose on Day 1
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: dupilumab — Solution for subcutaneous (SC) injection administration
  Other Names: DUPIXENT®; REGN668; SAR231893
  Arms: dupilumab
Drug: Placebo — Solution for SC injection administration
  Arms: Matching Placebo

SUMMARY:
The primary objective of the study is to assess the efficacy of dupilumab on skin lesions in patients with atopic hand and foot dermatitis.

The secondary objectives of the study are:

* To assess the efficacy of dupilumab on various other domains (pruritus, pain, sleep loss, health related QoL, work life impairment) in patients with atopic hand and foot dermatitis
* To evaluate the safety and tolerability of dupilumab administered to patients with atopic hand and foot dermatitis
* To evaluate systemic exposure and immunogenicity of dupilumab in patients with atopic hand and foot dermatitis

ELIGIBILITY:
Key Inclusion Criteria:

* Patients with involvement of at least 2 anatomical areas at screening and baseline
* Patients need to have an IGA hand and foot score of 3 or 4 (moderate-to-severe disease) at screening and baseline
* Patients with documented recent history (within 6 months before the screening visit) of inadequate response of atopic hand and foot dermatitis to topical medication(s)
* Patients meet the diagnosis criteria for atopic dermatitis (AD)
* Provide informed consent/assent signed by study patient or legally acceptable representative
* Patients need to have been compliant with the skin protection measures through the entire duration of the screening period

Key Exclusion Criteria:

* Treatment with dupilumab in the past
* Patients with a positive patch test reaction that are deemed to be clinically relevant as the current cause of the hand and foot dermatitis
* Patients with documented exposure to irritants believed to be a predominant cause of the current hand and foot dermatitis
* Treatment with systemic corticosteroids or non-steroidal immunosuppressive drugs within 4 weeks prior to baseline
* Known history of HIV/HBV/HCV infection
* Pregnant or breastfeeding women or planning to become pregnant or breastfeed during the patient's participation in this study
* Women of childbearing potential (WOCBP) who are unwilling to practice highly effective contraception prior to the initial dose/start of the first treatment and during the study

NOTE: Other protocol defined inclusion / exclusion criteria apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (42):
- United States (17):
  - Regeneron Study Site, Birmingham, Alabama
  - Regeneron Study Site, Redwood City, California
  - Regeneron Study Site, Washington D.C., District of Columbia
  - Regeneron Study Site, Macon, Georgia
  - Regeneron Study Site, Sandy Springs, Georgia
  - Regeneron Study Site, Columbus, Indiana
  - Regeneron Study Site, Rockville, Maryland
  - Regeneron Study Site, Saint Joseph, Missouri
  - Regeneron Study Site, St Louis, Missouri
  - Regeneron Study Site, Kew Gardens, New York
  - Regeneron Study Site, Mineola, New York
  - Regeneron Study Site, Winston-Salem, North Carolina
  - Regeneron Study Site, Portland, Oregon
  - Regeneron Study Site, Houston, Texas
  - Regeneron Study Site, Norfolk, Virginia
  - Regeneron Study Site, Morgantown, West Virginia
  - Regeneron Study Site, Milwaukee, Wisconsin
- Germany (11):
  - Regeneron Study Site, Langenau, Baden-Wurttemberg
  - Regeneron Study Site, Frankfurt am Main, Hesse
  - Regeneron Study Site, Augsburg
  - Regeneron Study Site, Berlin
  - Regeneron Study Site, Bonn
  - Regeneron Study Site, Dresden
  - Regeneron Study Site, Gera
  - Regeneron Study Site, Kiel
  - Regeneron Study Site, Lübeck
  - Regeneron Study Site, Mahlow
  - Regeneron Study Site, Münster
- Japan (7):
  - Regeneron Study Site, Kawasaki, Kanagawa
  - Regeneron Study Site, Sakai, Osaka
  - Regeneron Study Site, Shinjuku, Tokyo
  - Regeneron Study Site, Tachikawa, Tokyo
  - Regeneron Study Site, Kyoto
  - Regeneron Study Site, Osaka
  - Regeneron Study Site, Tokyo
- Poland (7):
  - Regeneron Study Site, Bialystok
  - Regeneron Study Site, Chorzów
  - Regeneron Study Site, Katowice
  - Regeneron Study Site, Kielce
  - Regeneron Study Site, Ostrowiec Świętokrzyski
  - Regeneron Study Site, Warsaw
  - Regeneron Study Site, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual anonymized participant data will be considered for sharing once the indication has been approved by a regulatory body, if there is legal authority to share the data and there is not a reasonable likelihood of participant re-identification.
Access Criteria: Qualified researchers may request access to anonymized patient level data or aggregate study data when Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc) for the product and indication, has the legal authority to share the data, and has made the study results publicly available (eg, scientific publication, scientific conference, clinical trial registry).
URL: https://vivli.org/

REFERENCES:
- [Derived] Cohen D, Bewley A, Wollenberg A, Hong HC, Armstrong A, Jonsen E, Maslin D, Thoning H, von Eyben R, Chovatiya R. Matching-Adjusted Indirect Comparison of the Efficacy of Delgocitinib Cream and Dupilumab in the Treatment of Moderate to Severe Atopic Hand Eczema. Dermatol Ther (Heidelb). 2025 Nov 15. doi: 10.1007/s13555-025-01592-y. Online ahead of print. PMID 41240207

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 170 participants were screened, 37 participants failed screening, and 133 participants were randomized. Of the 37 screen failures: 2 withdrew consent, 33 did not meet inclusion/exclusion criteria, 1 was lost to follow-up and 1 was for an unknown reason.
Groups:
- Matching Placebo: Administered subcutaneously (SC) once every 2 weeks (Q2W), following a loading dose on Day 1
- Dupilumab Q2W: Administered SC Q2W, following a loading dose on Day 1
Period: Overall Study
Arm/Group | Matching Placebo | Dupilumab Q2W
Started | 66 | 67
Completed | 53 | 60
Not Completed | 13 | 7
Not completed — Lost to Follow-up | 3 | 0
Not completed — Withdrawal by Subject | 7 | 6
Not completed — Lack of Efficacy | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Matching Placebo | Dupilumab Q2W | Total
Number analyzed (Participants) | 66 | 67 | 133
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.4 (14.66) | 35.8 (17.07) | 34.6 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 45 | 83
  Male | 28 | 22 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 63 | 64 | 127
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 53 | 53 | 106
  Black or African American | 4 | 3 | 7
  Asian | 8 | 9 | 17
  American Indian or Alaska Native | 0 | 1 | 1
  Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Hand and Foot Investigator Global Assessment (IGA) 0 or 1 at Week 16
Description: IGA is an assessment scale used to determine severity of hand and foot AD and clinical response to treatment on a 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Higher score is indicative of more severe disease.
Time Frame: At week 16
Measure: Number; unit: Percentage of participants
Arm/Group | Matching Placebo | Dupilumab Q2W
Number analyzed (Participants) | 66 | 67
Percentage of participants | 16.7 | 40.3
Statistical Analysis 1: Comparison: Matching Placebo vs Dupilumab Q2W; Test type: Superiority; p = 0.0030, Cochran-Mantel-Haenszel

2. Secondary Outcome: Percentage of Participants With Improvement (Reduction) of Weekly Average of Daily Hand and Foot Peak Pruritus Numerical Rating Scale (NRS) of ≥4 Points From Baseline to Week 16
Description: Pruritus NRS is an assessment tool that is used to report the intensity of a patient's pruritus (itch), both maximum and average intensity, during a 24-hour recall period; maximum itch intensity on a scale of 0 - 10 (0 = no itch; 10 = worst itch imaginable).
Time Frame: Baseline to week 16
Measure: Number; unit: Percentage of participants
Arm/Group | Matching Placebo | Dupilumab Q2W
Number analyzed (Participants) | 66 | 67
Percentage of participants | 13.6 | 52.2
Statistical Analysis 1: Comparison: Matching Placebo vs Dupilumab Q2W; Test type: Superiority; p < 0.0001, Mantel Haenszel; Difference = 38.6, 95% CI 2-sided [24.06 to 53.15]

3. Secondary Outcome: Percentage of Participants With Improvement (Reduction) of Weekly Average of Daily Hand and Foot Peak Pruritus NRS ≥3 From Baseline to Week 16
Description: as for outcome 2
Time Frame: Baseline to week 16
Measure: Number; unit: Percentage of participants
Arm/Group | Matching Placebo | Dupilumab Q2W
Number analyzed (Participants) | 66 | 67
Percentage of participants | 16.7 | 61.2

4. Secondary Outcome: Percent Change From Baseline to Week 16 in Weekly Average of Daily Hand and Foot Peak Pruritus NRS
Description: as for outcome 2
Time Frame: Baseline to week 16
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of change
Arm/Group | Matching Placebo | Dupilumab Q2W
Number analyzed (Participants) | 66 | 67
Percentage of change | -26.2 [-38.0 to -14.4] | -62.9 [-74.6 to -51.3]

5. Secondary Outcome: Percent Change in Modified Total Lesion Sign Score (mTLSS) for Hand/Foot Lesions From Baseline to Week 16
Description: mTLSS combines an evaluation of hand and foot eczema lesions severity; scores are summed, extending from a base estimation of 0 (no signs or symptoms) to the most extreme of 18 (more serious disease).
Time Frame: Baseline to Week 16
Population: The full analysis set (FAS) includes all randomized participants. Efficacy analyses will be based on the treatment allocated at randomization (as randomized).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of change
Arm/Group | Matching Placebo | Dupilumab Q2W
Number analyzed (Participants) | 66 | 67
Percentage of change | -31.0 [-42.6 to -19.4] | -69.4 [-80.9 to -58.0]

6. Secondary Outcome: Change From Baseline to Week 16 in Weekly Average of Daily Hand and Foot Peak Pain NRS
Description: Pain NRS Scale is an assessment tool used to report the intensity of a participant's pain. Participants will select the number between 0 and 10 that fits best to their worst pain intensity over the past 24 hours (0 = no pain and 10 = the worst pain possible).
Time Frame: Baseline to week 16
Population: The full analysis set (FAS) includes all randomized participants. Efficacy analyses will be based on the treatment allocated at randomization (as randomized). Here 'n' = number of evaluable participants at a specified point in time.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Matching Placebo | Dupilumab Q2W
Number analyzed (Participants) | 66 | 67
Score on a scale | -1.93 (0.432) | -4.66 (0.426)

7. Secondary Outcome: Mean Change From Baseline to Week 16 in Weekly Average of Daily Sleep NRS
Description: Sleep NRS is an 11-point scale (0 to 10) in which 0 indicates worst possible sleep while 10 indicates best possible sleep.
Time Frame: Baseline to week 16
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Matching Placebo | Dupilumab Q2W
Number analyzed (Participants) | 66 | 67
Score on a scale | -0.00 (0.335) | 0.88 (0.334)

8. Secondary Outcome: Change From Baseline to Week 16 in Percent Surface Area of Hand and Foot Involvement With Atopic Dermatitis (AD)
Time Frame: Baseline to week 16
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Percentage of hand and foot BSA
Arm/Group | Matching Placebo | Dupilumab Q2W
Number analyzed (Participants) | 66 | 67
Percentage of hand and foot BSA | -10.01 (2.388) | -16.70 (2.375)

9. Secondary Outcome: Percent Change From Baseline to Week 4 in Weekly Average of Daily Hand and Foot Peak Pruritus NRS
Description: Pruritus NRS is an assessment tool that is used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period; maximum itch intensity on a scale of 0 - 10 (0 = no itch; 10 = worst itch imaginable).
Time Frame: Baseline to week 4
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of change
Arm/Group | Matching Placebo | Dupilumab Q2W
Number analyzed (Participants) | 66 | 67
Percentage of change | -25.6 [-36.3 to -15.0] | -47.2 [-57.7 to -36.6]

10. Secondary Outcome: Percentage of Participants With Improvement (Reduction) of Weekly Average of Daily Hand and Foot Peak Pruritus NRS ≥4 From Baseline to Week 4
Description: as for outcome 9
Time Frame: Baseline to week 4
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Matching Placebo | Dupilumab Q2W
Number analyzed (Participants) | 66 | 67
Percentage of participants | 9.1 | 34.3

11. Secondary Outcome: Percent Change From Baseline to Week 16 in Hand Eczema Severity Index (HECSI) Score in Participants With Hand Dermatitis
Description: For participants with hand dermatitis HECSI is an instrument used in clinical trials to rate the severity of 6 clinical signs of hand eczema and the extent of the lesions on each of 5 hand areas by use of standard scales. The total HECSI score is based on a 4-point severity scale ranging from 0 (none/absent) to 3 (severe) and a 5-point scale rating the affected area(s) ranging from 0 (0% affected area) to 4 (76% to 100% affected area). The range for the combined HECSI score is from 0 to 360 (5x6x3x4).
Time Frame: Baseline to week 16
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Matching Placebo | Dupilumab Q2W
Number analyzed (Participants) | 65 | 64
Percentage of change | -33.8 (42.21) | -68.2 (25.56)

12. Secondary Outcome: Percentage of Participants With HECSI-75 at Week 16
Description: HECSI-75 is defined as HECSI score has ≥75% improvement from baseline for participants with hand dermatitis.
Time Frame: At week 16
Population: Efficacy analyses will be based on the treatment allocated at randomization (as randomized). Here 'n' = number of evaluable participants at a specified point in time.
Measure: Number; unit: Percentage of participants
Arm/Group | Matching Placebo | Dupilumab Q2W
Number analyzed (Participants) | 65 | 64
Percentage of participants | 21.5 | 46.9

13. Secondary Outcome: Percentage of Participants With HECSI-50 at Week 16
Description: HECSI-50 is defined as HECSI score has ≥50% improvement from baseline, for participants with hand dermatitis.
Time Frame: At week 16
Population: as for outcome 12
Measure: Number; unit: Percentage of participants
Arm/Group | Matching Placebo | Dupilumab Q2W
Number analyzed (Participants) | 65 | 64
Percentage of participants | 30.8 | 75.0

14. Secondary Outcome: Percentage of Participants With HECSI-90 at Week 16
Description: HECSI-90 is defined as HECSI score has ≥90% improvement from baseline for participants with hand dermatitis.
Time Frame: At week 16
Population: Efficacy analyses was based on the treatment allocated at randomization (as randomized). Here 'n' = number of evaluable participants at a specified point in time.
Measure: Number; unit: Percentage of participants
Arm/Group | Matching Placebo | Dupilumab Q2W
Number analyzed (Participants) | 65 | 64
Percentage of participants | 9.2 | 18.8

15. Secondary Outcome: Change From Baseline to Week 16 in Quality of Life in Hand Eczema Questionnaire (QOLHEQ)
Description: For participants with hand dermatitis, QOLHEQ is an instrument to assess disease specific Health Related Quality of Life (HRQOL) in those suffering from hand eczema. QOLHEQ overall scoring ranges as follows: 0 (best score) to 117 (worst score).
Time Frame: Baseline to week 16
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Matching Placebo | Dupilumab Q2W
Number analyzed (Participants) | 65 | 64
Score on a scale | -13.36 (21.222) | -38.70 (23.920)

16. Secondary Outcome: Mean Change From Baseline to Week 16 in Work Productivity and Impairment (WPAI) and Classroom Impairment Questionnaire (CIQ)
Description: WPAI + CIQ is a self-administered instrument used to capture the impairment to work productivity/classroom impairment and activity due to atopic hand and foot dermatitis. The WPAI+CIQ yields 4 types of scores: absenteeism, presenteeism, work/classroom productivity loss and activity impairment. All scores range from 0 to 100% with 100% indicating total work/classroom productivity impairment and 0 no impairment at all.
Time Frame: Baseline to week 16
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Matching Placebo | Dupilumab Q2W
Number analyzed (Participants) | 66 | 67
Score on a scale | -21.26 (3.761) | -36.39 (3.649)

17. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs) Through Week 16
Time Frame: Through week 16
Population: The safety analysis set (SAF) includes all randomized patients who receive at least one dose of study drug and will be analyzed as treated.
Measure: Number; unit: Percentage of participants
Arm/Group | Matching Placebo | Dupilumab Q2W
Number analyzed (Participants) | 66 | 67
Percentage of participants | 74.2 | 65.7

18. Secondary Outcome: Trough Concentration of Functional Dupilumab in Serum at Various Time Points
Time Frame: Up to week 28
Population: The pharmacokinetic analysis set (PKAS) includes all treated participants who received any amount of study drug (active or placebo [SAF]) and had at least 1 non-missing dupilumab measurement following the first dose of study drug or placebo. The PKAS is based on the actual treatment received (as treated) rather than as randomized. Here 'n' = number of evaluable participants at a specified point in time
Measure: Mean (Standard Deviation); unit: Milligrams per Liter (mg/L)
Groups:
- Dupilumab 300 mg - Adult Participants; Dupilumab 200 mg - Adolescent Participants; Dupilumab 300 mg - Adolescent Participants: Administered subcutaneously (SC) once every 2 weeks (Q2W), following a loading dose on Day 1
Arm/Group | Dupilumab 300 mg - Adult Participants | Dupilumab 200 mg - Adolescent Participants | Dupilumab 300 mg - Adolescent Participants
Number analyzed (Participants) | 49 | 6 | 6
Milligrams per Liter (mg/L)
  Week 0: number analyzed (Participants) | 43 | 6 | 6
  Week 0 | 0 (0) | 0 (0) | 0 (0)
  Week 16: number analyzed (Participants) | 48 | 6 | 4
  Week 16 | 51.2 (22.0) | 34.0 (10.7) | 37.1 (15.9)
  Week 28: number analyzed (Participants) | 43 | 2 | 5
  Week 28 | 7.37 (25.0) | 60.0 (84.9) | 7.54 (16.9)

19. Secondary Outcome: Number of Participants With Treatment-Emergent (TE) Anti-Drug Antibody (ADA)
Time Frame: Up to week 28
Population: The ADA analysis set (AAS) includes all treated participants who received any amount of study drug (active or placebo [safety analysis set]) and had at least one non-missing ADA result following the first dose of study drug or placebo. The ADA analysis set is based on the actual treatment received (active drug or placebo) rather than as randomized. Here 'n'= number of evaluable participants at a specified point in time.
Measure: Number; unit: Participants
Groups:
- Dupilumab Q2W: Administered subcutaneously (SC) once every 2 weeks (Q2W), following a loading dose on Day 1
Arm/Group | Matching Placebo | Dupilumab Q2W
Number analyzed (Participants) | 55 | 61
Participants
  Treatment-Boosted Response | 0 | 0
  Treatment-Emergent Response | 1 | 8

20. Secondary Outcome: Number of Participants With Treatment-Emergent ADA by Maximum Titer Category
Time Frame: Up to Week 28
Population: as for outcome 19
Measure: Number; unit: Participants
Arm/Group | Matching Placebo | Dupilumab Q2W
Number analyzed (Participants) | 55 | 61
Participants
  Low (<1,000) | 1 | 8
  Moderate (1,000 to 10,000) | 0 | 0
  High (>10,000) | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose to Week 28
Description: Participants included adults and adolescents (≥12 years) and were randomized at 1:1 to Dupilumab and placebo. For each group, adults and adolescents with body weight ≥60kg who had 300mg Q2W is similar to adolescents with body weight < 60kg who had 200mg Q2W. The 300mg Q2W and 200mg Q2W were similar dosing for participants with different weight and age, rather than different dosing for the same population. Thus, they were combined to compare Dupilumab with placebo.
Arm/Group | Matching Placebo | Dupilumab Q2W
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/67
Serious Adverse Events (participants affected / at risk) | 1/66 | 3/67
Other Adverse Events (participants affected / at risk) | 34/66 | 33/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Matching Placebo (N=66) | Dupilumab Q2W (N=67)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Matching Placebo (N=66) | Dupilumab Q2W (N=67)
COVID-19 (Infections and infestations) | 14 (14) | 11 (11)
Nasopharyngitis (Infections and infestations) | 8 (13) | 16 (18)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 7 (9)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 16 (18) | 6 (6)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2021-01-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT04417894/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-27): https://cdn.clinicaltrials.gov/large-docs/94/NCT04417894/SAP_001.pdf